CLINICAL TRIAL: NCT03991650
Title: REMOTE: Monitoring Telemedicine Platform in Patients With Anxiety Symptoms and Alcohol Use Disorder: Smartphone and Wearable Sensors
Brief Title: Monitoring Telemedicine Platform in Patients With Anxiety Symptoms and Alcohol Use Disorder
Acronym: REMOTE
Status: Completed | Type: Observational
Sponsor: humanITcare (Network)
Collaborators: Hospital Clinic of Barcelona (Other); European Institute of Innovation and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: humanITcare: Remote
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Anxiety Disorders; Alcohol Use Disorder; Depressive Disorder
Keywords: wearable; sensor; anxiety; monitoring; ehealth; Alcohol Use Disorder; depression
MeSH Terms: conditions — Anxiety Disorders; Alcoholism; Depressive Disorder; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: n=30 healthy participants will be recruited using social networks and leaflets of information distributed by the research team at the Hospital Cliníc de Barcelona.
  The participants will be monitored over the course of one month using the humanITcare app "U-Shine," which will track participant's sociability, device usage, and location frequency using mobile sensors. Participants' data will also be monitored with a FitBit device to track sleep schedules, heart rate, and step count. During the weekly follow-up, they will have to complete the three clinical questionnaires taken at the initial visit.
  Interventions: Behavioral: Monitoring with a device
- Experimental: The recruitment process will be carried out in patients of external consultations and the day hospital of the Addictions Unit at the Hospital Clinic of Barcelona.
  n=30 patients with Anxiety and Alcohol Use Disorder.
  The participants will be monitored over the course of one month using the humanITcare app "U-Shine," which will track participant's sociability, device usage, and location frequency using mobile sensors. Participants will also be monitored using a FitBit device to track sleep schedules, heart rate, and step count. During the weekly follow-up, they will have to complete the three clinical questionnaires taken at the initial visit.
  Interventions: Behavioral: Monitoring with a device

INTERVENTIONS:
Behavioral: Monitoring with a device — Participants will be monitored by an App.

SUMMARY:
The objective of this study is to analyze the physiological patterns of two groups of patients, one control and one with anxiety disorder and alcoholic abuse disorder using sensor data from mobile devices and wearables. This data will be compared to the data presented by three clinical questionnaires: State-trait Anxiety Inventory (STAI), the Alcohol Use Disorders Identification Test (AUDIT), and the Beck's Depression Inventory (BDI-II) in order to determine the feasibility of remote collected data.

DETAILED DESCRIPTION:
The objective of this study is to analyze the physiological patterns of two groups of patients, one control and one with anxiety disorder and alcoholic abuse disorder using sensor data from mobile devices and wearables. This data, collected by sensors, will be compared to the data presented by three clinical questionnaires: State-trait Anxiety Inventory (STAI), the Alcohol Use Disorders Identification Test (AUDIT), and the Beck's Depression Inventory (BDI-II) in order to determine the feasibility of using remote collected data in routine clinical practice. Furthermore, patient satisfaction with the app will be evaluated after the data collection phase.

This is a unicentric, case-controlled, longitudinal, evaluational, national study with two groups, one control of healthy individuals without symptoms of anxiety or depression, and another experimental group in which participants fulfill the given selection criteria for the trial. There are a total of 60 participants split evenly between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Alcohol use disorder (DSM 5) as main substance.
* Anxiety (STAI > percentile 33) and, if depressive symptoms, not clinically relevant as to accomplish DSM5 diagnostic criteria for mood disorders (major depressive disorder, bipolar disorder…).
* Having a mobile phone compatible with Android.
* Sign informed consent.

Exclusion Criteria:

* Mood disorder diagnoses (DSM5).
* Cognitive deficits that prevent the participation.
* Active intake of other substances (except for nicotine).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be a sample n = 60, with 30 healthy control subjects and 30 afflicted experimental subjects.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Self-reported Anxiety symptoms assessed with the State-Trait Anxiety Inventory (STAI) | One month, questionnaire taken 4 times (1/week)
  Taken through the application "Ushine". Participants receive STAI scores ranging from 0-60, 0 being lowest amount of symptoms, and 60 being the greatest amount of symptoms, which are then transformed into percentiles according to age and sex.
Sleep pattern | One month
  Monitoring of circadian rhythm using a motion sensor Fitbit and cardiac activity sensor
REM sleep time | One month
  monitoring of REM sleep patterns using a motion sensor Fitbit and cardiac activity sensor
Heart Rate | One month
  monitoring of heart rate using Fitbit sensor
Step count | One month
  Monitoring of daily step count using motion sensor FitBit
Distance travelled | One month
  Monitoring of distance travelled using GPS phone
Mobile device usage | One month
  Monitoring how often the patient's mobile device is used, determined by tracking the presence of a signal from their device
Sociability (number of incoming an outgoing calls and text messages) | One month
  The number of incoming and outgoing calls and text messages will be monitored using the UShine app algorithm
Change in Self-reported Depression symptoms assessed with the Beck's Depression Inventory (BDI-II) | One month, questionnaire taken 4 times (1/week)
  Taken through the application "Ushine". Participants receive BDI-II scores ranging from 1-63, with a score of 0-13 indicating minimal depression, 14-19 indicating mild depression, 20-28 indicating moderate depression, and 29-63 indicating severe depression.
Change in Self-reported Alcohol Abuse Symptoms assesed with the Alcohol Use Disorders Identification Test (AUDIT) | One month, questionnaire taken 4 times (1/week)
  Taken through the application "Ushine". Participants receive AUDIT scores ranging from 0-40. A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.

SECONDARY OUTCOMES:
Usability of the mobile application | One month
  Ease of usability of the mobile applications by participants will be scaled using the System Usability Scale (SUS). Final scores range from 0-100. A score of 51 or under means the system has serious faults in usability, a score of 68 means the system usability is about average, and a score of 80.3 or higher means the system usability is considered appreciable.
Satisfaction with the application | One month
  Participants' satisfaction with the Ushine application will be scaled using the Post-Study Usability Questionnaire (PSSUQ). Scores range from 0-100, 0 being least satisfactory and 100 being the most satisfactory. The PSSUQ has 3 sub-scores representing system usefulness, information quality, and interface quality, also scaled from 0-100. In all score sets, 0 is considered the least satisfactory and 100 is considered the most satisfactory.

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Gual, MD, Principal Investigator — Director of Addictions Unit. Hospital Clínic de Barcelona; Elsa Caballeria, Study Chair — Clinic Foundation for Biomedical Research; Hugo Lopez-Pelayo, MD, Study Chair — Addictions Unit, Hospital Clínic de Barcelona; Nuria Pastor Hernandez, MSc, Study Director — humanITcare, FollowHealth SL; Unai Sanchez Luque, MSc, Study Director — humanITcare, FollowHealth SL; Elizabeth Katayoun Khalilian, Study Chair — humanITcare, University of Texas at Austin
Locations (1):
- Hospitcal Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data sets that underlie results in the final study report will be available for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be available by the estimated date of September 2019, when study results are expected to be published
Access Criteria: Participants can access their own individual data records, only hospital researchers can access the aggregated data sets.

REFERENCES:
- [Background] Alonso J, Liu Z, Evans-Lacko S, Sadikova E, Sampson N, Chatterji S, Abdulmalik J, Aguilar-Gaxiola S, Al-Hamzawi A, Andrade LH, Bruffaerts R, Cardoso G, Cia A, Florescu S, de Girolamo G, Gureje O, Haro JM, He Y, de Jonge P, Karam EG, Kawakami N, Kovess-Masfety V, Lee S, Levinson D, Medina-Mora ME, Navarro-Mateu F, Pennell BE, Piazza M, Posada-Villa J, Ten Have M, Zarkov Z, Kessler RC, Thornicroft G; WHO World Mental Health Survey Collaborators. Treatment gap for anxiety disorders is global: Results of the World Mental Health Surveys in 21 countries. Depress Anxiety. 2018 Mar;35(3):195-208. doi: 10.1002/da.22711. Epub 2018 Jan 22. PMID 29356216
- [Background] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- [Background] Barrio P, Ortega L, Lopez H, Gual A. Self-management and Shared Decision-Making in Alcohol Dependence via a Mobile App: a Pilot Study. Int J Behav Med. 2017 Oct;24(5):722-727. doi: 10.1007/s12529-017-9643-6. PMID 28236288
- [Background] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- [Background] Reddy MS. Depression: the disorder and the burden. Indian J Psychol Med. 2010 Jan;32(1):1-2. doi: 10.4103/0253-7176.70510. No abstract available. PMID 21799550
- [Background] Menger V, Spruit M, Hagoort K, Scheepers F. Transitioning to a Data Driven Mental Health Practice: Collaborative Expert Sessions for Knowledge and Hypothesis Finding. Comput Math Methods Med. 2016;2016:9089321. doi: 10.1155/2016/9089321. Epub 2016 Aug 17. PMID 27630736
- [Background] Hsin H, Torous J, Roberts L. An Adjuvant Role for Mobile Health in Psychiatry. JAMA Psychiatry. 2016 Feb;73(2):103-4. doi: 10.1001/jamapsychiatry.2015.2839. No abstract available. PMID 26747695
- [Background] Insel TR. Digital Phenotyping: Technology for a New Science of Behavior. JAMA. 2017 Oct 3;318(13):1215-1216. doi: 10.1001/jama.2017.11295. No abstract available. PMID 28973224
- [Background] Bernert RA, Hom MA, Iwata NG, Joiner TE. Objectively Assessed Sleep Variability as an Acute Warning Sign of Suicidal Ideation in a Longitudinal Evaluation of Young Adults at High Suicide Risk. J Clin Psychiatry. 2017 Jun;78(6):e678-e687. doi: 10.4088/JCP.16m11193. PMID 28682534
- [Background] Bandelow B, Michaelis S. Epidemiology of anxiety disorders in the 21st century. Dialogues Clin Neurosci. 2015 Sep;17(3):327-35. doi: 10.31887/DCNS.2015.17.3/bbandelow. PMID 26487813
- [Background] Saeb S, Zhang M, Karr CJ, Schueller SM, Corden ME, Kording KP, Mohr DC. Mobile Phone Sensor Correlates of Depressive Symptom Severity in Daily-Life Behavior: An Exploratory Study. J Med Internet Res. 2015 Jul 15;17(7):e175. doi: 10.2196/jmir.4273. PMID 26180009
- [Background] Saeb S, Lattie EG, Kording KP, Mohr DC. Mobile Phone Detection of Semantic Location and Its Relationship to Depression and Anxiety. JMIR Mhealth Uhealth. 2017 Aug 10;5(8):e112. doi: 10.2196/mhealth.7297. PMID 28798010
- [Background] Sano A, Taylor S, McHill AW, Phillips AJ, Barger LK, Klerman E, Picard R. Identifying Objective Physiological Markers and Modifiable Behaviors for Self-Reported Stress and Mental Health Status Using Wearable Sensors and Mobile Phones: Observational Study. J Med Internet Res. 2018 Jun 8;20(6):e210. doi: 10.2196/jmir.9410. PMID 29884610
- [Background] Torous J, Staples P, Shanahan M, Lin C, Peck P, Keshavan M, Onnela JP. Utilizing a Personal Smartphone Custom App to Assess the Patient Health Questionnaire-9 (PHQ-9) Depressive Symptoms in Patients With Major Depressive Disorder. JMIR Ment Health. 2015 Mar 24;2(1):e8. doi: 10.2196/mental.3889. eCollection 2015 Jan-Mar. PMID 26543914
- [Background] Onnela JP, Rauch SL. Harnessing Smartphone-Based Digital Phenotyping to Enhance Behavioral and Mental Health. Neuropsychopharmacology. 2016 Jun;41(7):1691-6. doi: 10.1038/npp.2016.7. Epub 2016 Jan 28. No abstract available. PMID 26818126
- [Background] Trautmann S, Rehm J, Wittchen HU. The economic costs of mental disorders: Do our societies react appropriately to the burden of mental disorders? EMBO Rep. 2016 Sep;17(9):1245-9. doi: 10.15252/embr.201642951. Epub 2016 Aug 4. PMID 27491723
- [Background] Ghandeharioun, A., Fedor, S., Sangermano, L., Ionescu, D., Alpert, J., Dale, C., ... & Picard, R. (2017, October). Objective assessment of depressive symptoms with machine learning and wearable sensors data. In Affective Computing and Intelligent Interaction (ACII), 2017 Seventh International Conference on (pp. 325-332). IEEE.
- See also: World Health Organization. Global Status Report on Alcohol and Health (2018). — https://www.who.int/news-room/fact-sheets/detail/alcohol
- See also: World Health Organization. Mental depression and other common disorders: Global health estimates (2017). — https://apps.who.int/iris/bitstream/handle/10665/254610/WHO-MSD-MER-2017.2-eng.pdf